CLINICAL TRIAL: NCT00133627
Title: Safety and Efficacy Comparison Ketotifen Ophthalmic Solution in Patients With Seasonal Allergic Conjunctivitis
Brief Title: Ketotifen Ophthalmic Solution With Emedastine in Patients With Seasonal Allergic Conjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CZAD511ACN01
Record Dates: First submitted 2005-08-22; First posted 2005-08-23 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Seasonal Allergic Conjunctivitis
Keywords: Allergic; Conjunctivitis; Ketotifen; Histamine
MeSH Terms: conditions — Conjunctivitis | interventions — Ketotifen

INTERVENTIONS:
Drug: Ketotifen

SUMMARY:
Medications available for the treatment of seasonal allergic conjunctivitis include antihistamines. These medicines block the release of histamine, a substance in the body that is released when an allergic reaction occurs. Novartis (NVS) has developed an eye drop formulation of a well tried antihistamine called ketotifen. This study will compare the efficacy and the tolerability of ketotifen eye drops with emedastine, which is a popular treatment for seasonal allergic conjunctivitis in China.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 years or older.
* History of seasonal allergic conjunctivitis
* Presence of bilateral ocular itching/conjunctival hyperaemia (redness) at baseline:

  1. at least intensity degree 2 for itching, and
  2. at least intensity degree 4 for composite score of itching and conjunctival hyperaemia

Exclusion Criteria:

Other systemic/ophthalmic conditions

* Presence of any form of allergic conjunctivitis other than seasonal allergic conjunctivitis (e.g. perennial allergic conjunctivitis, vernal keratoconjunctivitis, atopic keratoconjunctivitis, giant papillary conjunctivitis).
* Active bacterial or viral conjunctivitis or history of ocular herpes.
* Presence or history of severe dry eye.

Previous treatments

* Any systemic or ocular corticosteroids within two (2) weeks prior to randomization.
* Any systemic or ocular mast cell stabilizers within two (2) weeks prior to randomization.
* Any other ophthalmic medication within three (3) days prior to randomization.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2005-04; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sun Xinghuai, Principal Investigator — Hospital of Shanghai Medical University
Locations (1):
- Hospital of Shanghai Medical University, Shanghai, China